CLINICAL TRIAL: NCT02761902
Title: Research to Characterize Normal Polysomnography Values in Healthy Children and Adolescents in China
Brief Title: Normal Polysomnography Values in Healthy Children and Adolescents in China
Acronym: PSGNV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Xin Ni, Hospital director, Beijing Children's Hospital
Other Study IDs: BCH-OSAHS-001
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Sleep Apnea
Keywords: Children; Polysomnography; sleep; obstructive sleep apnea;; Chinese
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Ecologic or Community
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Preschool group: 3-6 years old
- school age group: 7-12 years old
- Adolescence group: 13-15 years old

SUMMARY:
The study is designed to investigate normal polysomnographic respiratory values of Chinese healthy children and adolescents. By collecting the polysomnography (PSG) data and parameters of respiratory and sleep architecture，we hope to characterize normal polysomnography values in Chinese children and adolescents and to establish respiratory reference values for pediatric polysomnography which based on Chinese children's data.

DETAILED DESCRIPTION:
We plan to recruit 200 healthy, normal children and adolescents in this study, age ranging from 3 to 15 years. All of them will be invited to undergo an overnight polysomnography for at least 7h in Beijing Children's Sleep Center, meanwhile the parameters about sleep including EEG, electromyography, electrooculography, ECG, pulse oximetry arterial oxygen saturation (SpO2), chest wall and abdomen motion, oral and nasal airflow, and end-tidal PCO2 (PETCO2) will be recorded.

Based on the data we hope to give recommendation of normal PSG parameters of Chinese kids, and on this basis,to develop the diagnosis creteria for obstructive sleep apnea syndrome which will be more suitable for Chinese children conditions.

ELIGIBILITY:
Inclusion Criteria:

1.3 to 14-year-old children 2.from the community of China 3.healty children

Exclusion Criteria:

1. children with nocturnal snoring, continuous mouth breathing, difficulty breathing and apnea when sleep.
2. children with craniofacial abnormalities, such as Down's syndrome, Crouzon syndrome, achondroplasia, mandibular hypoplasia and facial mandibularetc hypoplasia.
3. children with history of upper respiratory tract infection nearly two weeks.
4. children with adenoids, tonsils, throat, glottis, trachea, lungs and history of thoracic surgery.
5. children with nose-sinusitis, allergic rhinitis, asthma, acut or purulent tonsillitis acute phase.
6. children with any medical or surgicaldiseases.
7. children who have to use use sedation to maintain sleep.
8. parents or child not understand the study or do not agree to take part in.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 3 to 14-year-old healthy children from the community of China
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
obstructive apneas per hour of sleep | 7 hours of sleep

SECONDARY OUTCOMES:
minimum oxygen desaturation of sleep | 7 hours of sleep
central apneas per hour of sleep | 7 hours of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Xin Ni, MD PHD, Study Director — Beijing Children's Hospital
Locations (1):
- Children's Sleep Center，Beijing,China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guilleminault C, Korobkin R, Winkle R. A review of 50 children with obstructive sleep apnea syndrome. Lung. 1981;159(5):275-87. doi: 10.1007/BF02713925. No abstract available. PMID 7300438
- [Background] Berry DT, Webb WB, Block AJ. Sleep apnea syndrome. A critical review of the apnea index as a diagnostic criterion. Chest. 1984 Oct;86(4):529-31. doi: 10.1378/chest.86.4.529. PMID 6478890
- [Background] Rosen CL, D'Andrea L, Haddad GG. Adult criteria for obstructive sleep apnea do not identify children with serious obstruction. Am Rev Respir Dis. 1992 Nov;146(5 Pt 1):1231-4. doi: 10.1164/ajrccm/146.5_Pt_1.1231. PMID 1443876
- [Background] Urschitz MS, Wolff J, Von Einem V, Urschitz-Duprat PM, Schlaud M, Poets CF. Reference values for nocturnal home pulse oximetry during sleep in primary school children. Chest. 2003 Jan;123(1):96-101. doi: 10.1378/chest.123.1.96. PMID 12527608
- [Background] Quan SF, Goodwin JL, Babar SI, Kaemingk KL, Enright PL, Rosen GM, Fregosi RF, Morgan WJ. Sleep architecture in normal Caucasian and Hispanic children aged 6-11 years recorded during unattended home polysomnography: experience from the Tucson Children's Assessment of Sleep Apnea Study (TuCASA). Sleep Med. 2003 Jan;4(1):13-9. doi: 10.1016/s1389-9457(02)00235-6. PMID 14592355
- [Background] Traeger N, Schultz B, Pollock AN, Mason T, Marcus CL, Arens R. Polysomnographic values in children 2-9 years old: additional data and review of the literature. Pediatr Pulmonol. 2005 Jul;40(1):22-30. doi: 10.1002/ppul.20236. PMID 15858805
- [Result] Uliel S, Tauman R, Greenfeld M, Sivan Y. Normal polysomnographic respiratory values in children and adolescents. Chest. 2004 Mar;125(3):872-8. doi: 10.1378/chest.125.3.872. PMID 15006944